CLINICAL TRIAL: NCT03220620
Title: Influence of Perioperative Fluid Therapy on Hemoglobin and Methemoglobin Levels in Major Abdominal Surgery
Brief Title: Influence of Perioperative Fluid Therapy on Hemoglobin and Methemoglobin Levels
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Thomas Mencke, Clinical Professor, University of Rostock
Other Study IDs: A 2017-0073
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Perioperative/Postoperative Complications; Fluid Overload; Hemoglobin H
Keywords: fluid therapy; perioperative; hemodilution
MeSH Terms: conditions — Postoperative Complications; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GDT Group: receives goal-directed therapy
  Interventions: Other: GDT
- Not GDT Group: receives no individualized goal-directed therapy

INTERVENTIONS:
Other: GDT — individualized fluid therapy
  Groups: GDT Group

SUMMARY:
The objective of the study is to evaluate influence of perioperative fluid therapy on Methemoglobin levels, and to changes in hemoglobin. Further, changes in Methemoglobin will be related to metabolic signs of oxidative stress (changes in blood lactate). Patients undergoing major abdominal surgery will be included into the study.

DETAILED DESCRIPTION:
Increasing plasma volume by intravenous administration of crystalloid and/or colloid solutions may cause a relative reduction in hemoglobin (Hb) concentration, a situation that is termed 'dilutional anemia'. Such hemodilution may lead to an iatrogenic reduction in oxygen-carrying capacity and the development of organ dysfunction. Paradoxically, large amounts of fluids that are administered with the aim of increasing oxygen delivery (DO2), as is frequently done as part of perioperative goal-directed therapy; this may lead to an actual decrease in the DO2 due to a decrease in Hb concentration.

Another potential parameter that may reflect the development of dilutional anemia is methemoglobin (MetHb), a form of Hb with reduced ability for oxygen binding. Experimental studies showed that dilutional anemia may lead to up-regulation of perivascular nitric oxide synthase (NOS) and increase NOS-derived nitric oxide (NO) leading to local vasodilation and oxidization of Hb to MetHb. MetHb may potentially serve as a biomarker of 'anemic stress' associated with reduced tissue perfusion during acute hemodilution.

ELIGIBILITY:
Inclusion Criteria:

* major abdominal surgery
* informed consent

Exclusion Criteria:

* violation of study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Influence of perioperative fluid therapy on hemoglobin levels | during surgery
  Influence of perioperative fluid therapy on hemoglobin levels
Influence of perioperative fluid therapy on Methemoglobin levels | during surgery
  Influence of perioperative fluid therapy on Methemoglobin levels

SECONDARY OUTCOMES:
Influence of perioperative fluid therapy on changes in lactate | during surgery
  Influence of perioperative fluid therapy on changes in lactate
Influence of perioperative fluid therapy on SvO2 | during surgery
  Influence of perioperative fluid therapy on SvO2

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mencke, Prof., Principal Investigator — University of Rostock
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No